CLINICAL TRIAL: NCT03663855
Title: Effect of Increasing Doses of Tiopronin on Cystine Capacity in Patients With Cystinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00642
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria | interventions — Tiopronin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cystinuria Patients (Experimental)
  Interventions: Drug: Tiopronin

INTERVENTIONS:
Drug: Tiopronin — Phase 1: No medication, Phase 2: 500mg PO daily x 7 days (total 500mg), Phase 3: 500mg PO BID x 7 days (total 1g), Phase 4: 1g PO BID x 7 days (total 2g)

SUMMARY:
The purpose of this study is to determine the minimum effective dose of the cysteine binding thiol drug (CBTD) Tiopronin on urine cystine capacity, which is a measure of cystine solubility in the urine, in patients with cystinuria to evaluate the effect of escalating doses of cystine binding thiol drugs on the cystine capacity of the urine. The overall goal will be to help guide therapy and ultimately minimize unnecessary side effects caused by larger dosages.

Cystinuria is a rare genetic disease that can lead to significant morbidity in affected patients due to the recurrent nature of the disease. This study will follow the levels of urine cystine capacity in order to help guide treatment and to use lower than usually prescribed Tiopronin doses to decrease the potential side effects while maintaining therapeutic benefit. This will increase adherence with the medications by decreasing the burden of the large number of pills that need to be taken daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed laboratory diagnosis of cystinuria who meet the following criteria: (1) stone analysis demonstrating cystine as a component, or (2) increased urinary cystine excretion (>250mg/24hrs in adults).
* A medical regimen that includes Tiopronin.
* Willing to use a medically accepted form of birth control, if female and of child bearing- potential
* Ability to reliably urinate in a collection vessel and measure urine volume.
* Ability to give informed consent.
* Documentation of a stable complete blood count (CBC) and urinalysis (UA) in the six month period prior to the date of enrollment.
* Enrollment in Rare Kidney Stone Consortium (RKSC) Protocol 6401 (Cystinuria Registry)

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or trying to become pregnant
* Patients with renal colic
* Patients who are scheduled to undergo a surgical procedure
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification. Researchers who provide a methodologically sound proposal.
Supporting Information: CSR, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Multiple efforts to contact the PI/study team for the relevant data have failed. Therefore, per sequence data are not available to be reported for this assessment.
Groups:
- Cystinuria Patients: Phase 1: No medication, Phase 2: 500mg PO daily x 7 days (total 500mg), Phase 3: 500mg PO BID x 7 days (total 1g), Phase 4: 1g PO BID x 7 days (total 2g)
Period: Overall Study
Arm/Group | Cystinuria Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Multiple efforts to contact the PI/study team for the relevant data have failed. Therefore, per intervention data are not available to be reported for this assessment.
Arm/Group | Cystinuria Patients
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cystine Capacity From Baseline
Description: This measure reflects the ability of urine to take up more cystine
Time Frame: Baseline; Day 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cystinuria Patients
Number analyzed (Participants) | 10
mg/L
  Phase 1 | -63.6 (24.8)
  Phase 2 | 76 (18.1)
  Phase 3 | 53.4 (17.7)
  Phase 4 | 103.1 (27.4)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Multiple efforts to contact the PI/study team for the relevant data have failed. Therefore, per dose level data are not available to be reported for this assessment.
Arm/Group | Cystinuria Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03663855/Prot_SAP_000.pdf